CLINICAL TRIAL: NCT00382616
Title: Studying the Effects of Phosphatidylserine Enriched With Omega-3 Fatty Acids on Symptoms of Attention-Deficit/Hyperactivity Disorder in Children
Brief Title: Supplementation of Phosphatidylserine (PS) and n-3 Long Chain Fatty Acids (EPA, DHA) in Children With ADHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TASMC-03-NV-220-CTIL
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Last update posted 2006-11-07 (Estimated); Status verified 2006-09

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
Keywords: behavioral problems; learning problems; inattentive; impulsive; hyperactive; children; phosphatidylserine; long-chain polyunsaturated fatty acid; eicosapentaenoic acid; docosahexaenoic acid; omega3:omega6 ratio; eicosapentaenoic acid:arachidonic acid ratio; Test of Variables of Attention; ADHD index scores
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Problem Behavior; Impulsive Behavior; Spasm

INTERVENTIONS:
Drug: Phosphatidylserine-Omega3

SUMMARY:
To determine whether supplementation of omega-3 long-chain polyunsaturated fatty acid conjugated to phosphatidylserine rather than triglycerides (fish oil) could affect Attention-deficit/hyperactivity disorder symptoms in children.

DETAILED DESCRIPTION:
BACKGROUND Attention-deficit/hyperactivity disorder (ADHD) encompasses a broad constellation of behavioral and learning problems, clinically describes inattentive, impulsive, and/or hyperactive children. These patients are characterized by low blood LC-PUFA (LC-PUFA) levels; however the LC-PUFA supplementation effect on ADHD symptoms is not clear.

METHODS Eighty-three ADHD children (3:1 boys:girls), 8-13 years old, were assigned in a randomized, double-blind, placebo-controlled parallel design to receive 250 mg/d of eicosapentaenoic acid + docosahexaenoic acid provided as phosphatidylserine (300 mg/d PS-Omega3), or fish oil or placebo for 3 months. Stimulant medication or other dietary supplements were prohibited. The measured outcomes were inattention and impulsivity, evaluated by Test of Variables of Attention (TOVA) and blood lipids profile.

ELIGIBILITY:
Inclusion Criteria:

* 8 and 13 years of age; diagnosed as having ADHD; otherwise healthy;

Exclusion Criteria:

* significant sensory or neurological limitations, epilepsy, mental retardation, psychosis, or pervasive developmental disorder; medications with known central nervous system effects such as tranquilizers, antidepressants, stimulants (including methylphenidate and amphetamines), sedating antihistamines and some asthma medications and dietary supplements but vitamins

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90
Dates: Start 2004-07; Study Completion 2005-01

PRIMARY OUTCOMES:
Laboratory assessment of inattention and impulsivity with Test of Variables of Attention (TOVA)
Blood lipids profile

SECONDARY OUTCOMES:
Hebrew translation of Conners' Parent Rating Scale-Revised, Short Form
Hebrew translation of the Child Behavior Checklist for Age 4-18, Parent form by Achenbach

CONTACTS AND LOCATIONS:
Overall Officials: Nachum Vaisman, MD, Principal Investigator — Clinical Nutrition Unit, Sourasky Tel Aviv Medical Center
Locations (1):
- Clinical Nutrition Unit, Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Derived] Vaisman N, Kaysar N, Zaruk-Adasha Y, Pelled D, Brichon G, Zwingelstein G, Bodennec J. Correlation between changes in blood fatty acid composition and visual sustained attention performance in children with inattention: effect of dietary n-3 fatty acids containing phospholipids. Am J Clin Nutr. 2008 May;87(5):1170-80. doi: 10.1093/ajcn/87.5.1170. PMID 18469236